CLINICAL TRIAL: NCT05366140
Title: Prospective Follow-up of Patients Undergoing Instrumented Thoracic and Lumbar Arthrodesis Supplemented by the Implanet Jazz System TM.
Brief Title: Thoracic-Lumbar Arthrodesis- Implanet Jazz
Status: Recruiting | Type: Observational
Sponsor: Francis Farhadi (Other)
Collaborators: Implanet America, Inc. (Unknown)
Responsible Party: Sponsor-Investigator, Francis Farhadi, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Other Study IDs: 73811
Record Dates: First submitted 2022-05-04; First posted 2022-05-09 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Spondylolisthesis; Spinal Stenosis; Degenerative Disease
Keywords: Thoracic-Lumbar Arthrodesis; Spinal fusion; back pain
MeSH Terms: conditions — Spondylolisthesis; Spinal Stenosis; Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Prospective follow-up of patients who have received instrumented lumbar arthrodesis supplemented the Implanet Jazz System(TM) — To assess the clinical outcomes of patients receiving standard of care Implanet Jazz System(TM) at the time of their instrumented lumbar arthrodesis.

SUMMARY:
Establish a data repository of patients who have undergone single, two-, or three-level lumbar instrumented arthrodesis procedures supplemented by the Implanet Jazz System.

DETAILED DESCRIPTION:
To collect and organize data into a repository from the Principal Investigator's and other Site Investigators' patients who are undergoing single, two-level, or three-level lumbar instrumented arthrodesis procedures supplemented by the Implanet Jazz SystemTM at participating centers. This device is designed to provide a stable interface between spinal constructs and the rods; it can be secured around vertebral structures (such as the lamina, transverse or spinous processes) from T1 to L5 and is intended to provide temporary stabilization as a bone anchor during the development of a solid body fusion. Of note, these patients will receive the supplemental support of the Implanet Jazz Sublaminar Band as their clinical standard of care deems necessary and separately from study participation.

Clinical data will be collected as indicated at 6 weeks, as well as 3, 6, 12, 24, 36, 48, and 60 months post-operatively in the database.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, 18 years of age and older
* Qualified candidate for hybrid thoracolumbar fixation with the Implanet Jazz System TM during arthrodesis surgery.

Exclusion Criteria:

* Individuals who have not yet reached the age of 18.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult men and women of any/all ethnic groups who are appropriate candidates for hybrid thoracolumbar fixation and will receive the Implanet Jazz System (TM) during their arthrodesis surgery.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-02-03 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
clinical prospective review- Prospective Database study for future studies | 5- years
  Collecting clinical measurements. Examples of these clinical measurements are the VAS Pain Scale, SF-36, NDI, and ODI.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No